CLINICAL TRIAL: NCT07295795
Title: Blood Sampling Pre- and Post-Propofol to Characterize the Blood Proteome Using Different Research Assays
Brief Title: Blood Sampling Pre- and Post-Propofol Administration to Characterize the Blood Proteome Using Different Research Assays
Status: Not yet recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10002371; 002371-CC
Record Dates: First submitted 2025-12-19; First posted 2025-12-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-18

CONDITIONS: Critically Ill Surgical Patients
Keywords: Propofol; Blood Proteome; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill surgical patients: Participant consented for a surgical procedure (primary surgical protocol) anticipated to require induction with propofol.

SUMMARY:
Background:

Propofol is a drug that helps people fall asleep quickly and stay asleep during surgery, so they do not feel any pain. This drug is also used to sedate critically ill people who must be on a ventilator (a machine to help them breathe). To better understand how to interpret blood tests in these ill people, researchers need to know more about how the drug itself may change proteins in the blood.

Objective:

To collect blood samples from people before and after propofol is administered for surgery.

Eligibility:

People aged 18 years or older who are scheduled for surgery that requires sedation with propofol.

Design:

Participants will have data collected. This data will include age, sex, and ethnicity. They will be asked about their medical history.

Participants will have blood samples collected before and after they receive propofol for their surgery. The blood will be collected from lines already installed for the surgery; no new needlesticks will be done for the study. A total of 3 teaspoons of blood will be drawn.

The samples will be compared to each other to look for any changes caused by the drug.

No follow-up visits are required.

DETAILED DESCRIPTION:
Study Description:

This is a blood procurement research protocol. The study will collect a total of 3 blood samples at 2 timepoints (1 blood sample prior to propofol and 2 after propofol dosing) from up to 10 participants pre- and post-induction of anesthesia with propofol to characterize the effects of propofol on the measurement of the blood proteome using different research assays. Blood samples will be withdrawn from existing intravenous access so that no additional interventions are required. The PI, or team designee, will have a discussion with the primary surgeon to determine suitability of the potential participant for eligibility. If determined suitable, the participant will be recruited by invitation. All potential participants will be consented to a primary surgical protocol; consent to this protocol will be secondary and obtained prior to the procedure.

Objectives:

Primary Objective:

The primary objective of this research protocol is to procure blood samples from participants prior to and post propofol administration to quantify the impact of propofol on the quantification of the blood proteome.

Endpoints:

The primary endpoint of this study is the reproducibility measurements based on the repeated quantifications of biomarkers using different biomarker assays Pre- and Post-Propofol administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Participant consented for a surgical procedure (primary surgical protocol) anticipated to require induction with propofol.
3. Male or female aged 18 years or older.
4. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Surgical procedure not utilizing propofol
2. Hemoglobin < 7 ug/dL at the time of enrollment
3. Inability to sign consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant consented for a surgical procedure (primary surgical protocol) anticipated to require induction with propofol. Male or female aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the reproducibility measurements based on the repeated quantifications of biomarkers using different biomarkers assays pre- and post-propofol. | 1 year
  The investigators would like to use the O-link Explore HT and SomaScan Discovery v4.1assay on samples from participants who are critically ill. In order to do this understanding, the impact of propofol on each analyte must be understood as there is potential for interference with propofol in each sample.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Mannes, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002371-CC.html